CLINICAL TRIAL: NCT02491619
Title: Correlation Between Buccolingual Dental Inclination and Bone Thickness After Orthodontic Decompensation in Patients With Class III Dentofacial Deformities
Brief Title: Correlation Between Dental Inclination and Bone Thickness in Patients With Class III Dentofacial Deformities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michelle Sendyk (Other)
Responsible Party: Sponsor-Investigator, Michelle Sendyk, Master degree student, University of Sao Paulo
Organization: University of Sao Paulo (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: sendyk001
Record Dates: First submitted 2015-06-24; First posted 2015-07-08 (Estimated); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Dentofacial Deformities
Keywords: Angle class III; tomography; tooth inclination; bone thickness
MeSH Terms: conditions — Dentofacial Deformities; Malocclusion, Angle Class III

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Orthodontic decompensation (Experimental): Orthodontic decompensation in patients with class III dentofacial deformities
  Interventions: Procedure: orthodontic decompensation

INTERVENTIONS:
Procedure: orthodontic decompensation — Evaluation of the correlation between bone thickness and tooth inclination previously and after orthodontic treatment of decompensation due to orthognathic surgery

SUMMARY:
The correlation between tooth inclination and bone thickness and the comparison between thickness measurements and buccolingual inclination before and after dental decompensation will be evaluated through tridimensional images in individuals with class III dentofacial deformities.

DETAILED DESCRIPTION:
Class III dentofacial deformity is associated with important functional, psychological and aesthetic changes and thus individuals affected by this type of deformity are motivated in seeking treatment. The sample will consist of three-dimensional images of 40 individuals with Class III dentofacial deformities. From these images generated by CBCT scans, the buccolingual inclinations of all teeth and maxillo-mandibular alveolar bone thickness in three different heights will be measured (3, 6 and 8 mm) from the cementoenamel junction through the Dolphin 3D® program. The 3D scans of the sample will be evaluated in two stages: the initial stage and after dental decompensation at the end of pre-surgical orthodontic phase. Pearson correlation test will be used to verify the relationship between tooth inclination and bone thickness. The thickness measurements and buccolingual inclination will be compared between treatment times (initial and pre-surgical) using paired Student t-test.

ELIGIBILITY:
Inclusion Criteria:

* Brazilian nationality;
* Class III malocclusion, for molars and canines;
* Concave facial profile;
* Indications for orthodontic-surgical treatment;
* Craniofacial growth finalized ;
* Absence of tooth extractions;
* No local and / or general contraindications for surgery;
* No previous orthodontic-surgical treatment;
* Good dental and periodontal conditions.

Exclusion Criteria:

* Facial asymmetry;
* Absence of teeth (except the third molars);
* Periodontal disease and vertical or horizontal bone resorption;
* Extensive metal restorations;
* Previous orthodontic treatment;
* Root anomalies.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in tooth inclination and bone thickness after tooth decompensation | 12 months after the begginning of orthodontic treatment, prior to orthognathic surgery

CONTACTS AND LOCATIONS:
Overall Officials: José Rino Neto, PhD, Study Chair — University of Sao Paulo
Locations (1):
- University of Sao Paulo, São Paulo, São Paulo, Brazil